CLINICAL TRIAL: NCT02711748
Title: Can Medical Personnel Properly Proceed in the Case of a Patient With Bradycardia?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Łukasz Szarpak, Lukasz Szarpak, Medical University of Warsaw
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 02.012.1MR
Record Dates: First submitted 2016-02-22; First posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bradycardia (Experimental): Treatment In case of bradycardia. The patient unconscious, breathing preserved in ECG - bradycardia 40 / min with pulse.
  Interventions: Device: electrostimulation
- PEA (Experimental): In case of bradycardia. The patient unconscious, not breathing, the ECG - bradycardia 30 / min - no pulse. Pulseless electrical activity
  Interventions: Device: cardiopulmonary resuscitation

INTERVENTIONS:
Device: electrostimulation — Electrostimulation using manual defibrillator
  Arms: Bradycardia
Device: cardiopulmonary resuscitation — CPR according to guidelines of European Resuscitation Council. Cardiopulmonary resuscitation using manual defibrillator
  Arms: PEA

SUMMARY:
The study aims to assess the regularity of the proceedings in the case of a patient with bradycardia ECG.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* maximum 1 year of work experience in medicine
* paramedics, nurses, physicians

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Questionnaire to assess effectiveness of the rhythm recognition and participants' knowledge on life-threatening rhythms | intraoperative
  The effectiveness of the rhythm recognition. participants knowledge on life-threatening rhythms

SECONDARY OUTCOMES:
Time to take proper action | intraoperative
  time from rhythm interpretation to proper conduct

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Department of Emergency Medicine, Warsaw, Masovia, Poland

IPD SHARING:
Plan to Share IPD: Undecided